CLINICAL TRIAL: NCT03902457
Title: Histomorphometric and Cone Beam Computed Tomography Assessments on the Influence a Collagen Membrane Placed Subjacent the Sinus Mucosa After Maxillary Sinus Floor Augmentation. A Randomized Clinical Trial.
Brief Title: Histomorphometric and Tomographic Assessment on the Influence of the Placement of a Collagen Membrane Subjacent the Sinus Mucosa After Maxillary Sinus Floor Augmentation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ARDEC Academy (Network)
Collaborators: Corporacion Universitaria Rafael Nunez (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CBCT sinus membrane
Record Dates: First submitted 2019-03-30; First posted 2019-04-04 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-09

CONDITIONS: Alveolar Bone Loss
Keywords: maxillary sinus; collagen membrane; CBCT; Histology
MeSH Terms: conditions — Alveolar Bone Loss | interventions — Sinus Floor Augmentation

STUDY DESIGN:
Intervention Model Description: Clinical trial
Who Masked: Care Provider, Investigator
Masking Description: An author not involved in the surgeries will perform the randomization process. The assignments will be sealed within opaque envelopes that will be opened after the completion of the elevation of the sinus mucosa.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- test site (Experimental): The sinus mucosa will be elevated and, at the test sites, a collagen membrane will be placed subjacent the sinus mucosa
  Interventions: Procedure: Maxillary sinus augmentation
- control site (Experimental): The sinus mucosa will be elevated and, at the control sites, a collagen membrane will not be placed subjacent the sinus mucosa
  Interventions: Procedure: Maxillary sinus augmentation

INTERVENTIONS:
Procedure: Maxillary sinus augmentation — Maxillary sinus augmentation procedures have become increasingly popular procedures before placement of dental implants in posterior maxillae that have suffered severe bone loss due to sinus pneumatization, alveolar bone atrophy, or trauma.
  Other Names: maxillary sinus lift, maxillary sinus elevation

SUMMARY:
the purpose of the study is to look for differences in dimensional variations of augmented maxillary sinuses with or without the placement of a collagen membrane subjacent the sinus mucosa.

DETAILED DESCRIPTION:
Material and Methods: After the elevation of the maxillary sinus mucosa, a collagen membrane with standard dimensions will be placed at the test sites subjacent the sinus mucosa and the elevated space will be filled with a xenograft, both test and control groups. A collagen membrane will be placed to cover the antrostomy at both groups and sutures will be provided to close the wound. After six months of healing, mini-implants will be installed. After 9 months, biopsies containing the mini-implants will be harvested for histomorphometric analyses. CBCTs will be taken for all patients before surgery (T0), after 1 week from sinus floor augmentation (T1) and after 9 months of healing (T2). Osseointegration of the mini-implants and dimensional changes over time of soft and hard tissues will be evaluated on the CBCTs.

ELIGIBILITY:
Inclusion Criteria:

* presence of an edentulous atrophic zone in the posterior segment of the maxilla
* height of the sinus floor ≤4 mm
* desiring a prosthetic restoration of the zone using a fix prosthesis supported by implants;
* ≥ 21 years of age
* good general health
* no contraindication for oral surgical procedures
* not being pregnant

Exclusion Criteria:

* present a systemic disordered
* had a chemotherapic or radiotherapeutic treatment
* are smokers >10 cigarettes per day
* have an acute or a chronic sinusitis
* had a previous bone augmentation procedures in the zone of interest.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-02-03 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Changing in height of the elevated zone | The CBCTs will be taken before surgery (T0) and 1-week (T1) and 9 months (T2) after surgery.
  Measurements will be assessed in the medial, middle and lateral regions of the elevated zone using the cone beam computerized tomographies (CBCTs) taken in various periods.
New bone-to-implant contact | Mini-implants will be installed six months after sinus lifting and retrieved after three months of healing.
  Measurements will be assessed between the most coronal (B) and the most apical (A) contacts of new bone to the implant surface.

SECONDARY OUTCOMES:
Changing in mucosa thickness | The CBCTs will be taken before surgery (T0) and 1-week (T1) and 9 months (T2) after surgery.
  Measurements will be assessed in the cone beam computerized tomographies (CBCTs) taken in various periods. Comparisons among the CBCTs of each participants will be performed.
New bone density around the mini-implant, from B to A and up to a distance of 400 µm from the implant surface. | Mini-implants will be installed six months after sinus lifting and retrieved after three months of healing
  Measurements will be assessed using a point counting procedure, superposing a lattice with squares of 50 µm over the histological image.

CONTACTS AND LOCATIONS:
Locations (1):
- Colombia, Cartagena, Cartagena, Colombia

IPD SHARING:
Plan to Share IPD: Yes
the results will be published in a Journal
Supporting Information: CSR
Time Frame: will be become available after the time required by the journal for publication and will be available all the time the journal is active.

REFERENCES:
- [Result] Schwartz-Arad D, Herzberg R, Dolev E. The prevalence of surgical complications of the sinus graft procedure and their impact on implant survival. J Periodontol. 2004 Apr;75(4):511-6. doi: 10.1902/jop.2004.75.4.511. PMID 15152813
- [Result] Nolan PJ, Freeman K, Kraut RA. Correlation between Schneiderian membrane perforation and sinus lift graft outcome: a retrospective evaluation of 359 augmented sinus. J Oral Maxillofac Surg. 2014 Jan;72(1):47-52. doi: 10.1016/j.joms.2013.07.020. Epub 2013 Sep 24. PMID 24071378
- [Result] Kawakami S, Lang NP, Iida T, Ferri M, Apaza Alccayhuaman KA, Botticelli D. Influence of the position of the antrostomy in sinus floor elevation assessed with cone-beam computed tomography: A randomized clinical trial. J Investig Clin Dent. 2018 Nov;9(4):e12362. doi: 10.1111/jicd.12362. Epub 2018 Aug 24. PMID 30144303
- [Result] Kawakami S, Lang NP, Ferri M, Apaza Alccayhuaman KA, Botticelli D. Influence of the height of the antrostomy in sinus floor elevation assessed by cone beam computed tomography- a randomized clinical trial. Int J Oral Maxillofac Implants. 2019 January/February;34(1):223-232. doi: 10.11607/jomi.7112. Epub 2018 Dec 5. PMID 30521653
- [Result] Iida T, Carneiro Martins Neto E, Botticelli D, Apaza Alccayhuaman KA, Lang NP, Xavier SP. Influence of a collagen membrane positioned subjacent the sinus mucosa following the elevation of the maxillary sinus. A histomorphometric study in rabbits. Clin Oral Implants Res. 2017 Dec;28(12):1567-1576. doi: 10.1111/clr.13027. Epub 2017 Jun 7. PMID 28593727
- [Result] Omori Y, Ricardo Silva E, Botticelli D, Apaza Alccayhuaman KA, Lang NP, Xavier SP. Reposition of the bone plate over the antrostomy in maxillary sinus augmentation: A histomorphometric study in rabbits. Clin Oral Implants Res. 2018 Aug;29(8):821-834. doi: 10.1111/clr.13292. Epub 2018 Jun 7. PMID 29876969
- [Result] Aimetti M, Romagnoli R, Ricci G, Massei G. Maxillary sinus elevation: the effect of macrolacerations and microlacerations of the sinus membrane as determined by endoscopy. Int J Periodontics Restorative Dent. 2001 Dec;21(6):581-9. PMID 11794569
- [Result] Khoury F. Augmentation of the sinus floor with mandibular bone block and simultaneous implantation: a 6-year clinical investigation. Int J Oral Maxillofac Implants. 1999 Jul-Aug;14(4):557-64. PMID 10453672
- [Result] Lundgren S, Andersson S, Gualini F, Sennerby L. Bone reformation with sinus membrane elevation: a new surgical technique for maxillary sinus floor augmentation. Clin Implant Dent Relat Res. 2004;6(3):165-73. PMID 15726851
- [Result] Choi BH, Zhu SJ, Jung JH, Lee SH, Huh JY. The use of autologous fibrin glue for closing sinus membrane perforations during sinus lifts. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2006 Feb;101(2):150-4. doi: 10.1016/j.tripleo.2005.04.008. Epub 2005 Sep 19. PMID 16448914
- [Result] Pikos MA. Maxillary sinus membrane repair: report of a technique for large perforations. Implant Dent. 1999;8(1):29-34. doi: 10.1097/00008505-199901000-00003. PMID 10356454
- [Result] Proussaefs P, Lozada J. The "Loma Linda pouch": a technique for repairing the perforated sinus membrane. Int J Periodontics Restorative Dent. 2003 Dec;23(6):593-7. PMID 14703763
- [Result] Proussaefs P, Lozada J, Kim J. Effects of sealing the perforated sinus membrane with a resorbable collagen membrane: a pilot study in humans. J Oral Implantol. 2003;29(5):235-41. doi: 10.1563/1548-1336(2003)0292.3.CO;2. PMID 14620686
- [Result] Testori T, Wallace SS, Del Fabbro M, Taschieri S, Trisi P, Capelli M, Weinstein RL. Repair of large sinus membrane perforations using stabilized collagen barrier membranes: surgical techniques with histologic and radiographic evidence of success. Int J Periodontics Restorative Dent. 2008 Feb;28(1):9-17. PMID 18351198
- [Result] Kim YK, Yun PY, Oh JS, Kim SG. Prognosis of closure of large sinus membrane perforations using pedicled buccal fat pads and a resorbable collagen membrane: case series study. J Korean Assoc Oral Maxillofac Surg. 2014 Aug;40(4):188-94. doi: 10.5125/jkaoms.2014.40.4.188. Epub 2014 Aug 26. PMID 25247149
- [Result] Scala A, Lang NP, Velez JU, Favero R, Bengazi F, Botticelli D. Effects of a collagen membrane positioned between augmentation material and the sinus mucosa in the elevation of the maxillary sinus floor. An experimental study in sheep. Clin Oral Implants Res. 2016 Nov;27(11):1454-1461. doi: 10.1111/clr.12762. Epub 2016 Jan 11. PMID 26754150
- [Result] Favero V, Lang NP, Canullo L, Urbizo Velez J, Bengazi F, Botticelli D. Sinus floor elevation outcomes following perforation of the Schneiderian membrane. An experimental study in sheep. Clin Oral Implants Res. 2016 Feb;27(2):233-40. doi: 10.1111/clr.12576. Epub 2015 Feb 25. PMID 25712609
- [Result] Zijderveld SA, Schulten EA, Aartman IH, ten Bruggenkate CM. Long-term changes in graft height after maxillary sinus floor elevation with different grafting materials: radiographic evaluation with a minimum follow-up of 4.5 years. Clin Oral Implants Res. 2009 Jul;20(7):691-700. doi: 10.1111/j.1600-0501.2008.01697.x. PMID 19453567

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-04-04): https://cdn.clinicaltrials.gov/large-docs/57/NCT03902457/Prot_SAP_001.pdf